CLINICAL TRIAL: NCT01978028
Title: Differential Gene Expression in Patients With Heart Failure and Iron Deficiency - Effects of Ferric Carboxymaltose
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vifor-HF
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ferric carboxymaltose (Active Comparator): ferric carboxymaltose
  Interventions: Drug: ferric carboxymaltose
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ferric carboxymaltose
  Arms: ferric carboxymaltose
Drug: placebo
  Arms: placebo

SUMMARY:
The primary efficacy objective of this study is to evaluate the effect of ferric carboxymaltose on mitochondrial gene activation pattern after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure of New York Heart Association Class II or III, a left ventricular ejection fraction of ≤ 40% for patients in NYHA class II or ≤ 45% for patients in NYHA class III, a hemoglobin level at the screening visit between 9.5-13.5 g/dl, and iron deficiency, which is defined as serum ferritin level < 100µg/l or between 100 and 299 µg/l, when transferring saturation is < 20%.
* Age ≥18 years
* Obtained informed consent
* Stable pharmacological therapy during the last 4 weeks (with the exception of diuretics)

Exclusion Criteria:

* Hemochromatosis, iron overload, defined as TSAT > 45%
* Known hypersensitivity to Ferinject®.
* Known active infection, CRP>20 mg/L, clinically significant bleeding, active malignancy.
* Chronic liver disease and/or screening alanine transaminase (ALT) or aspartate transaminase (AST) above three times the upper limit of the normal range.
* Immunosuppressive therapy or renal dialysis (current or planned within the next 6 months).
* History of erythropoietin, i. v. or oral iron therapy, and blood transfusion in previous 12 weeks and/or such therapy planned within the next 6 months.
* Unstable angina pectoris as judged by the investigator, clinically significant uncorrected valvular disease or left ventricular outflow obstruction, obstructive cardiomyopathy, poorly controlled fast atrial fibrillation or flutter, poorly controlled symptomatic brady- or tachyarrhythmias.
* Acute myocardial infarction or acute coronary syndrome, transient ischemic attack or stroke within the last 3 months.
* Coronary-artery bypass graft, percutaneous intervention (e.g. cardiac, cerebrovascular, aortic; diagnostic catheters are allowed) or major surgery, including thoracic and cardiac surgery, within the last 3 months.
* Participation in a CHF training program.
* Known HIV/AIDS.
* Inability to fully comprehend and/or perform study procedures in the investigator's opinion.
* Vitamin B12 and/or serum folate deficiency according to the laboratory (re-screening is possible after substitution therapy).
* Pregnancy or lactation.
* Participation in another clinical trial within previous 30 days and/or anticipated participation in another trial during this study.
* Anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The primary efficacy objective of this study is to evaluate the effect of ferric carboxymaltose on mitochondrial gene activation pattern after 12 weeks of treatment | 12 weeks
  The primary efficacy objective of this study is to evaluate the effect of ferric carboxymaltose on mitochondrial gene activation pattern after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frank Enseleit, MD, Principal Investigator — University Hospital Zurich, Devision of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No